CLINICAL TRIAL: NCT00180856
Title: A Phase II Study of Radiofrequency Ablation of Lung Tumors
Brief Title: Radiofrequency Ablation of Lung Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFPULM
Record Dates: First submitted 2005-09-11; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer; Metastasis
Keywords: Lung metastasis; Lung cancer; Radiofrequency ablation
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis | interventions — Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation

SUMMARY:
Radiofrequency ablation has achieved impressive results in the treatment of unresectable primary and metastatic liver cancer. Animal studies have demonstrated that radiofrequency can fully ablate lung tumors in animal models. We set up a prospective study to evaluate the local efficacy of radiofrequency ablation of lung neoplasms. The aim of the study is to prospectively evaluate local efficacy with a minimal follow-up of one year, tolerance, lung disease-free survival and survival after radiofrequency ablation of lung tumors (primary lung cancer or lung metastases).

DETAILED DESCRIPTION:
Radiofrequency (RF) ablation has achieved impressive results in the treatment of unresectable primary and metastatic liver cancer. Animal studies have demonstrated that RF can fully ablate lung tumors in animal models. We set up a prospective study to evaluate the local efficacy of radiofrequency ablation of lung neoplasms with a minimal follow-up of one year. The primary endpoint was to determine the rate of incomplete local treatment at 1 year. The secondary endpoints were to evaluate tolerance, survival, disease-free survival and lung tumor-free survival. Patients are followed-up by CT scan examination at day 1 or 2 before discharge from the hospital, then at 2, 4, 6, 9 and 12 months and then at 2 years

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral unresectable primary or metastatic lung tumors <= 40 mm and a number of tumor <=5
* Tumors located more than 1 cm from the hilum, and not involving soft tissues or mediastinum.
* Malignancy histologically proven for pulmonary nodules in patients with no history of cancer outside the lung.
* Lung tumors in patients with a known distant cancer history, has to be either histologically proven or a demonstrated change in size of at least 25% in their largest diameter is required on CT during the previous year
* Pretreatment imaging work-up within 4 weeks of scheduled RF ablation (at least a chest CT and an abdomino-pelvic CT)
* If a tumor is found outside the lung, it has to be amenable to complete eradication with RF or RF plus surgery
* Lung spirometry within 4 weeks of treatment with a FEV1 >= 1 liter
* Written informed consent.

Exclusion Criteria:

* Uncorrectable coagulopathy with a prothrombin time greater than 1.5 and a platelet count below 106/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01

PRIMARY OUTCOMES:
Incomplete local treatment

SECONDARY OUTCOMES:
Survival
Lung disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Thierry De Baere, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Jean Pallussière, MD, Principal Investigator — Institut Bergonié
Locations (2):
- France (2):
  - Institut Bergonié, Bordeaux
  - Institut Gustave Roussy, Villejuif